CLINICAL TRIAL: NCT05261113
Title: Clinical Study to Evaluate the CE-IOUS Outcome-relevant Impact on the Surgical Treatment of Liver Tumours and Liver Metastases
Brief Title: CE-IOUS Impact on Surgical Strategy of Liver Tumours and Liver Metastases
Status: Completed | Type: Observational
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Florian Bitterer, Principal Investigator, University of Regensburg
Other Study IDs: 17-699-101
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Liver Neoplasms; Liver/Hepatobiliary Cancer; Colorectal Cancer Metastatic; Metastases; Surgery; Ultrasound
Keywords: CE-IOUS; IOUS
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention cohort: Patients that were operated due to liver neoplasms with use of CE-IOUS
  Interventions: Procedure: CE-IOUS
- Control cohort: Patients that were operated due to liver neoplasms without use of CE-IOUS

INTERVENTIONS:
Procedure: CE-IOUS — Use of contrast-enhanced intraoperative ultrasound during liver surgery
  Groups: Intervention cohort

SUMMARY:
Contrast-enhanced intraoperative ultrasound (CE-IOUS) plays an increasingly important role in the surgical therapy planning of primary liver lesions as well as liver metastases.

The present study was designed to evaluate the significance of CE-IOUS by specificity and sensitivity and particularly the impact it exerts on the surgical strategy.

A secondary aim was assessing the outcome relevance of surgeries influenced by CE-IOUS.

DETAILED DESCRIPTION:
CE-IOUS has been used during hepatobiliary surgery for almost 25 years. During this time, it has proven to be an excellent diagnostic tool for detecting and characterising previously unknown lesions.

It is still unclear to what extent the findings of this imaging modality impacts the strategy of such operations.

The currently planned study is intended to evaluate the impact of contrast-enhanced intraoperative ultrasound on the surgical procedure in hepatic surgery.

For this purpose, patient data of the time period between 2017 and 2019 was prospectively analysed.

Another aim of the study was to measure the outcome relevance of CE-IOUS. This assessment was carried out by comparing an intervention cohort with a control cohort. The control cohort consisted of patients that were operated due similar liver lesions as the intervention cohort however did not receive CE-IOUS during the operation. Aspects like the recurrence free time and overall survival rate of the two cohorts were compared together with the patients' characteristics of the groups themselves.

ELIGIBILITY:
Inclusion Criteria:

* Operations during study period from 01/2017 until 12/2019
* Elective liver surgery in the department of surgery at the University Hospital Regensburg
* Liver resections due to primary hepatic tumours (benign, malignant) or hepatic metastases
* Liver surgery with intraoperative use of CE-IOUS

Exclusion Criteria:

* Intraoperative use of CE-IOUS outside the department of surgery
* Liver transplantations
* Use of CE-IOUS only for exclusion of hepatic metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that received elective liver surgery in the study centre during the study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Impact on surgical strategy during CE-IOUS | 01.01.2017 - 31.12.2019
  Frequency of surgeries changed due to findings of CE-IOUS together with histopathological correlation.
Outcome relevance of CE-IOUS | 01.01.2017 - 30.06.2021
  Comparison of recurrence-free interval, overall survival rate of the intervention cohort and control cohort as well as the groups themselves.

SECONDARY OUTCOMES:
Sensitivity and Specificity of CE-IOUS compared to other imaging methods | 01.01.2017 - 31.12.2019
  Accuracy of CE-IOUS in comparison to CT and MRI measured right localisation as well as classification of tumour dignity.

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Schlitt, MD Prof., Study Chair — Head of Department
Locations (1):
- University Hospital Department of Surgery, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided